CLINICAL TRIAL: NCT03748966
Title: Calcitriol Monotherapy for X-Linked Hypophosphatemia: Effects on Mineral Ions, Growth and Skeletal Parameters
Brief Title: Calcitriol Monotherapy for X-Linked Hypophosphatemia
Status: Active, not recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Collaborators: National Institute of Arthritis and Musculoskeletal and Skin Diseases (NIAMS) (NIH)
Responsible Party: Principal Investigator, Eva Liu, Assistant Professor of Medicine, Massachusetts General Hospital
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2016P001000
Record Dates: First submitted 2018-11-19; First posted 2018-11-21 (Actual); Last update posted 2025-10-01 (Actual); Status verified 2025-09

CONDITIONS: X-linked Hypophosphatemia; Hypophosphatemic Rickets; Hypophosphatemic Rickets, X-Linked Dominant
Keywords: XLH; calcitriol; x-linked hypophosphatemia; rickets; 1,25 dihydroxyvitamin D; bone disorder; rare bone disease; vitamin D; hypophosphatemic rickets
MeSH Terms: conditions — Familial Hypophosphatemic Rickets; Rickets, Hypophosphatemic; Rickets; Bone Diseases | interventions — Calcitriol; 1,25-dihydroxyvitamin D

STUDY DESIGN:
Intervention Model Description: Adults or children (age 3-17) with X-linked hypophosphatemia (XLH) will be enrolled the study. All research subjects will be treated with optimized doses of calcitriol alone (without phosphate supplementation) for one year.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Adults with XLH (Experimental): Adults with X-linked hypophosphatemia will be treated with optimized doses of calcitriol (without phosphate supplementation) for one year
  Interventions: Drug: Calcitriol
- Children with XLH (Experimental): Children (age 3-17) with X-linked hypophosphatemia will be treated with optimized doses of calcitriol (without phosphate supplementation) for one year
  Interventions: Drug: Calcitriol

INTERVENTIONS:
Drug: Calcitriol — Adults and children (age 3-17) with X-linked hypophosphatemia will be treated with calcitriol therapy without phosphate supplementation. Doses of calcitriol will be escalated and optimized in the first three months of the study. Calcitriol is an oral medication taken once a day.
  Other Names: 1,25 dihydroxyvitamin D

SUMMARY:
Children and adults with XLH recruited will be treated with calcitriol alone (without phosphate supplementation) for one year, during which the calcitriol dose will be escalated during the first 3 months of therapy. The investigators hypothesize that treatment of adults and children with XLH alone will improve serum phosphate levels and skeletal mineralization without causing an increase in kidney calcifications. The study will also examine if calcitriol therapy will improve growth in children.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of XLH with family history excluding male-to-male transmission, or positive genotype for PHEX mutation
* Serum PTH levels less than 1.5x the upper limit of normal
* Serum calcium levels less than 10.0 mg/dl
* eGFR >= 60 mL/min/1.73m2
* 25(OH) vitamin D level >= 20 ng/dL

Exclusion Criteria:

* Known allergy to calcitriol
* Pregnancy or breast feeding
* Use of skeletally active agents such as bisphosphonates, teriparatide, SERMS, hormone replacement therapy and progesterone-only contraceptive agents (combination oral contraceptive use in premenopausal women is not an exclusion criterion).
* Unwilling or unable to stop therapy with calcitriol and phosphate therapy for two weeks prior to study
* Therapy with cinacalcet within the past two weeks
* Current use of growth hormone therapy
* Use of diuretics or medications that alter renal handling of mineral ions.
* Use of glucocorticoids for more than 14 days in the past 12 months with the exception of inhaled agents.
* History of malignancy except basal and squamous cell carcinoma of the skin.
* Significant history of psychiatric disease per DSM-5.
* Substance use disorder per DSM-5.
* Significant cardiopulmonary disease (unstable CAD or stage D ACC/AHA heart failure).
* Absence of laboratory values for serum calcium, phosphate and creatinine in the 24 months prior to enrollment.

Ages: 3 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2019-03-28 (Actual); Primary Completion 2025-03-01 (Actual); Study Completion 2026-05 (Estimated)

PRIMARY OUTCOMES:
Change from baseline in serum phosphate in adults and children with XLH | up to 12 months
Change from baseline in TmP/GFR in adults and children with XLH | up to 12 months
  a measure of kidney resorption of phosphate
Rickets score for children with XLH | up to 12 months
  a score of rickets severity determined by reading x-rays of wrists and knees (10 point Thacher score with 0 being normal and 10 being severe)
Change from baseline in nephrocalcinosis grade | up to 12 months
  determine if there is change in amount of calcifications in the kidneys: graded from grade 0 (normal) to grade IV (stone formation, solitary focus of echos at the tip of the renal pyramid)

SECONDARY OUTCOMES:
Growth in children with XLH | up to 12 months
  Z-score of growth

CONTACTS AND LOCATIONS:
Overall Officials: Eva Liu, MD, Principal Investigator — Massachusetts General Hospital and Brigham and Women's Hospital
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Liu ES, Martins JS, Raimann A, Chae BT, Brooks DJ, Jorgetti V, Bouxsein ML, Demay MB. 1,25-Dihydroxyvitamin D Alone Improves Skeletal Growth, Microarchitecture, and Strength in a Murine Model of XLH, Despite Enhanced FGF23 Expression. J Bone Miner Res. 2016 May;31(5):929-39. doi: 10.1002/jbmr.2783. Epub 2016 Feb 2. PMID 26751835